CLINICAL TRIAL: NCT05726214
Title: Effectiveness of the Fragicare Exercise Program on Functional and Socio-sanitary Management Parameters
Brief Title: Exercise Program for Maintaining Physical Function and Frailty on Dwelling Older Adults
Acronym: FragiCare
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties with the recruitment process
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, Ana Rodriguez Larrad, Associate profesor, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: FragiCare exercise program
Record Dates: First submitted 2023-01-25; First posted 2023-02-13 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Frailty
Keywords: exercise; physical activity; funcionality; elderly; dwelling; socio-sanitary management
MeSH Terms: conditions — Frailty; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Due to the difficulties observed during the recruitment, an allocation based on participants' will was conducted to ensure attendance. Thus, participants were allocated by convenience into two groups
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): The control group received general recommendations for maintaining physically active and reducing sedentary behaviors. This was done verbally and through written material.
  Interventions: Other: Recommendations for active lifestyle
- Intervention Group (Experimental): The intervention group received the same recommendations as the control group. In addition, they participated in a multicomponent physical exercise program consisting of a) 1 face-to-face weekly multicomponent session (Rodriguez-Larrad et al. BMC Geriatrics (2017)), and b) 2 autonomous sessions at home following the Vivifrail program. Our targeted duration of 24 weeks was missed due to the lack of predisposition expressed by some participants, once the recruitment was completed, to continue during summer vacation. Therefore, the intervention was restructured to be carried out in 16 weeks.
  Face-to-face supervised sessions lasted 1 hour and included strength, balance, and flexibility exercises (50%-75% of the 1 repetition maximum for strength exercises). The volume, intensity and difficulty of the exercises were individualized based on the initial performance of each participant, and progressed as the participants' physical capacity evolved.
  Interventions: Other: Exercise; Other: Recommendations for active lifestyle

INTERVENTIONS:
Other: Exercise — The face-to-face multicomponent program entailed:
  * Strength training of upper and lower limbs. Familiarization phase included 2-3 exercises of 1-2 series and 8-12 repetitions per session. During the acquisition phase, 2-3 exercises of 2-3 series and 8-12 repetitions at a higher velocity. The resting time between sets lasted 1-3 minutes.
  * Balance exercises included proprioception, agility and weight transfer exercises. Difficulty progressively increased by reducing the base of support, by including multidirectional displacements, walking on tiptoe or heels, body-weight transfer, dynamic exercises modifying the centre of gravity, and stressing postural muscles and by sensorial reductions.
  * Flexibility exercises: Static stretching maintained during 20-30s carried out at the end of each session.
  The Vivifrail exercise wheel corresponding to each participant was given according to their functional level type.
  Arms: Intervention Group
Other: Recommendations for active lifestyle — After the baseline assessments, all participants received individualized counseling for following physically active lifestyle and reducing sedentary behaviors. Participants were encouraged to increase the physical activity time and intensity, and to hourly break the sedentary time while at home. The recommendations were transmitted verbally and through written material.

SUMMARY:
Older people living in their homes and receiving social assistance are at a high risk of suffering functional loss, hospitalization and/or developing disability. This condition is known as frailty. Exercise programs including strength, balance and flexibility training have demonstrated to prevent, delay or even treat frailty. However, participation in this type of exercise programs is very limited in the group of older adults mentioned above.

The present study seeks to evaluate the effects of an exercise program designed to maintain or improve physical function and frailty. The hypothesis is that people who participate in the physical exercise program will maintain or improve their physical capacity, their frailty and psycho-affective status, their quality of life, and generate a lower demand for social and health services compared to those people who do not exercise.

DETAILED DESCRIPTION:
Frailty is recognized as a syndrome that encompasses a high risk of suffering functional loss, hospitalization and/or developing dependency, among other adverse health events. It is considered a modifiable factor, capable of being reversed if intervention is made in the early stages of its development. The implementation of multicomponent physical exercise programs has been proven to prevent, delay or even treat frailty. However, participation in this type of exercise programs is very limited in older people living in their homes and receiving social assistance. Social assistance in Spain is recognized as a care and preventive nature service intended to help older adults in a situation of dependency, or risk of dependency, to remain at their homes, offering them the required domestic and personalized assistance that enables their development in their own homes and their integration into the community environment, avoiding situations of isolation. Older people living in their homes and receiving social assistance population is characterized by being particularly vulnerable, since it presents high rates of frail people that are in the initial stages of dependency, which makes them a target to significantly benefit from the effects of exercise.

The approach to tackling frailty has become a Public Health priority at a European, state and regional level, as it affects both the health and social systems in an increasingly aging society. Nevertheless, there are currently no frailty management models in an integrated manner between health and social service systems. In this context arises the FRAGICARE project, which aspires to develop a model of shared health and social management, sustainable in the long term, which promotes the permanence of the older adults in their usual social environment, respecting their lifestyles and preferences. This model is supported by a digital platform uploaded in the cellular, fed by the data collected by the professionals who are in charge of the home care service provided to the dwelling older adults. In the event of a significant change in the conditions that affect these older adults (fall, reduction in functional level, modification of the nutritional pattern, change in the social network, ...), the platform generates a series of alarms that are referred to their healthcare and/or social professional, who will reassess and, if necessary, adjust the care plan. These alarms have been defined by a multidisciplinary group of experts and piloted in a previous project. In this way, the model seeks to provide individualized, continuous and coordinated care between the basic social services system and the health system (primary and specialized care services).

The objective of the present study is to assess the effects of a physical exercise program from a multidimensional perspective, including physical function, frailty status, psycho-affective parameters, and quality of life. In addition, we will also evaluate the effect of the program in the number of alarms generated by the digital platform to the social and health services.

The hypothesis is that people who participate in the physical exercise program will maintain or improve their physical function, their frailty status, psycho-affective capacity, quality of life, and generate a lower number of social and health services alarms compared to those people who do not exercise.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or older.
* Home care users managed by the municipal social network.
* In a stable situation (no worsening, no convalescence, no hospital discharge).
* Frail or pre-frail individuals.

Exclusion Criteria:

* At the end of life.
* <60 on the Barthel Index.
* Cognitive impairment that affects their decision-making ability (Mini Mental State Examination, MMSE <24).
* Subjects that, on Home Care Service's assistant's criteria, do not meet the conditions to be included in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline Short Physical Performance Battery (SPPB) total score at 4 months | Baseline and 4 months
  The SPPB consists of three tasks that evaluate the lower extremities' function: balance, walking speed and sit-to-stand 5 times from a chair. In each task 0 to 4 points can be scored, to obtain a total score between 0 and 12 points. Higher values indicate better function.

SECONDARY OUTCOMES:
Change from baseline Fried's frailty phenotype score at 4 months | Baseline and 6 months
  Frailty was analyzed with the 5 criteria suggested by Fried: unintentional weight loss, weakness or poor handgrip strength, self-reported exhaustion, slow walking speed, and low physical activity. The presence of each criterion scored with one point, the total score ranging between 0-5 points. A higher score indicates higher frailty.
Change from baseline height at 4 months | Baseline and 4 months
  Height was measured and reported in meters, following ISAK's criteria.
Change from baseline weight at 4 months | Baseline and 4 months
  Weight was measured and reported in kilograms, following ISAK's criteria.
Change from baseline hand grip at 4 months | Baseline and 4 months
  The grip strength of each hand was measured with a manual dynamometer. This variable is related to the general strength of the subject, where higher values indicate greater strength.
Change from baseline Eight Foot up and Go (8-FUG) at 4 months | Baseline and 4 months
  The test measures the time the subject needs to stand from a chair, walk 8 feet (2,5 meters), turn around, get back to the chair, and sit. The longer the time to complete the test, the worse the performance. Leaning on the thighs or the chair is allowed to stand.
Change from baseline Nutritional state at 4 months | Baseline and 4 months
  The nutritional state was evaluated using the short form (SF) of the Mini-Nutritional Assessment (MNA). The score of SF-MNA oscillates between 0 and 14. The nutritional state can be classified as normal nutrition (12 to 14 points), potential risk of malnutrition (8 to 11 points), and malnutrition (<7 points).
Change from baseline Cognition at 4 months | Baseline and 4 months
  The Montreal Cognitive Assessment was used to evaluate the cognitive function of participants. It analyzes the following abilities: attention, concentration, executive functions (including abstraction ability), memory, language, visual-construction-related abilities, calculus, and orientation. The maximum score is 30 points; a score of 26 or higher is considered normal.
Change from baseline Anxiety and Depression at 4 months | Baseline and 4 months
  Anxiety and Depression Goldberg Scale. The scale is formed of two subscales with nine questions each: the anxiety subscale and the depression subscale. The total score in both subscales goes from 0 to 9, since each question scores 1 point if the answer is affirmative, and 0 points if it is not. In the anxiety subscale, the cut-off point which determines that the participant has a risk of suffering anxiety is 4 points or more, and the depression risk is 2 points or more. In both subscales the higher the score, the higher the risk.
Change from baseline health-related quality of life at 4 months | Baseline and 4 months
  European Quality of Life-5 Dimensions (EQ-5D) questionnaire. Participants will self-rate their health on a vertical visual analogue scale (score range: 0-100), where the endpoints are labeled 'The worst health you can imagine' and 'The best health you can imagine'. Higher values indicate better quality of life.
Change from baseline Meaning in Life Questionnaire score at 4 months | Baseline and 4 months
  The Spanish version of the Meaning in Life Questionnaire was used. It contains 10 questions that evaluate the meaning of life. The questionnaire has Likert-type options which go from "absolutely false", which scores 1 point, to "absolutely true", which scores 7 points. The total score goes from 10 to 70 points. Higher scores indicate better values.
Change from baseline Satisfaction With Life Scale score at 4 months | Baseline and 4 months
  It is a 5-question scale with Likert-type answers of 5 categories that examines de global grade of satisfaction with life. Possible answers go from absolutely untrue (1) to absolutely true (5). A score of 5 to 25 points can be obtained. Higher values indicate better satisfaction with life.
Change from baseline Subjective Happiness Scale score at 4 months | Baseline and 4 months
  The scale consists of 4 questions. The first three questions include 7 possible Likert-type answers, where the minimum score is 1 (little happy) and the maximum is 7 (totally happy). In the last question, the Likert scale is modified, where the minimum score is 1 (not at all) and the maximum is 7 (a great deal). The maximum score possible is 28 points. Higher values indicate a better score.
Sociodemographic information | Baseline and in any moment that any of them might change (place of residence, cohabitation model and social network) up to 4 months.
  Date of birth, sex, place of residence, cohabitation model and social network. Any change in those circumstances will be recorded from baseline assessment up to 4 months.
Number of falls | From baseline assessment up to 4 months
  The number of falls each participant suffered during the program was recorded on a self-reported basis and from Home Care Service's registers. It also included the number of falls in the last 4 months from the Home Care Service's registers.
  This was prospectively recorded from the date of baseline assessment until the date of the first documented fall, assessed up to 4 months.
Attendance to the face-to-face exercise sessions | From the first session up to the last one during the 4 months
  The number of face-to-face sessions carried out by each participant was collected by the trainer in each session.
Attendance to the autonomous sessions at home | From the first session up to the last one during the 4 months
  The number of completed autonomous sessions at home was self-reported. Participants registered them on a sheet, which was delivered weekly to the trainer during the program.
Alarms to the social and health care services | Daily from baseline assessment up to 4 months
  Professionals in charge of the home care service provided to the dwelling older adults collected data in a digital platform regarding the health and social conditions of the person they care for. In the event of a significant change in the conditions that affected the older adults (fall, reduction in functional level, modification of the nutritional pattern, change in the social network, ...), the platform generated a series of alarms. These alarms were then referred to the older adult health and/or social care professionals. We assessed the number of alarms referred to the health and/or social care professionals of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Ana AR Rodriguez Larrad, Principal Investigator — UPV/EHU
Locations (1):
- University of the Basque Country, Leioa, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared under reasonable demand
Supporting Information: CSR
Time Frame: When data will be collected and analyzed
Access Criteria: Data will be shared under reasonable demand to the principal investigator

REFERENCES:
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Stewart A, Marfell-Jones M, International Society for Advancement of Kinanthropometry. International Standards for Anthropometric Assessment. ISAK, 2011
- [Background] Mayordomo MM. Análisis Dinamométrico de la Mano: Valores Normativos en la Población Española. Madrid: Universidad Complutense de Madrid, Servicio de Publicaciones,; 2011
- [Background] Rikli, R.E., Jones, C.J., 2001. Senior Fitness Test. Champaign: Human Kinetics. (ISBN 0-7360-3356-3364
- [Background] Kaiser MJ, Bauer JM, Ramsch C, Uter W, Guigoz Y, Cederholm T, Thomas DR, Anthony P, Charlton KE, Maggio M, Tsai AC, Grathwohl D, Vellas B, Sieber CC; MNA-International Group. Validation of the Mini Nutritional Assessment short-form (MNA-SF): a practical tool for identification of nutritional status. J Nutr Health Aging. 2009 Nov;13(9):782-8. doi: 10.1007/s12603-009-0214-7. PMID 19812868
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Goldberg D, Bridges K, Duncan-Jones P, Grayson D. Detecting anxiety and depression in general medical settings. BMJ. 1988 Oct 8;297(6653):897-9. doi: 10.1136/bmj.297.6653.897. PMID 3140969
- [Background] Steger MF, Frazier P, Kaler M, Oishi S. The meaning in life questionnaire: Assessing the presence of and search for meaning in life. J Couns Psychol. 2006;53(1):80-93
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Extremera N, Fernández-Berrocal P. The Subjective Happiness Scale: Translation and Preliminary Psychometric Evaluation of a Spanish Version. Soc Indic Res. 2014;119:473-481.